CLINICAL TRIAL: NCT03322644
Title: Development and Feasibility Testing of an Internet-based Pain Self-management Program for Persons With Acute Recurrent and Chronic Pancreatitis Pain (The IMPACT Study)
Brief Title: Internet-based Pain Self-management for Persons With Acute Recurrent and Chronic Pancreatitis Pain
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Mayo Clinic (Other); University of Pittsburgh Medical Center (Other); Ohio State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mayo IRB #17-007214; U01DK108334 (NIH)
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Pancreatitis, Chronic; Pancreatitis, Acute Recurrent
Keywords: Pancreatitis; Pain; Internet Intervention; Behavioral Intervention
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based CBT intervention (Experimental): In addition to standard medical care, participants in the Internet-based CBT group will receive access to the Pancreatitis Pain Course and will be asked to complete all online modules over 2 months using their own smartphone or computer. A coach will guide participants through the weekly lessons.
  Interventions: Behavioral: Internet-based CBT intervention
- Wait list control group (No Intervention): Participants assigned to the Wait list control group will be asked to continue with any recommendations made by their clinic provider and will not be offered any internet-based content until after they complete the 5 month assessments (i.e. Months 5-7).

INTERVENTIONS:
Behavioral: Internet-based CBT intervention — The Internet-delivered Pancreatitis Pain Course consists of 5 lessons: 1) introduction, education, and symptom identification, 2) thought monitoring and challenging, 3) controlled breathing and pleasant activity scheduling, 4) activity pacing, and 5) relapse prevention and goal setting. Participants aim to complete one online lesson weekly for 5 weeks, and have up to 2 months to complete the course. Each lesson has a homework assignment to encourage participants to practice and apply skills. A coach who is part of the Seattle Children's Research Institute study team will make weekly contact with participants in the intervention arm through telephone or secure e-mail, for a period of between 10-15 minutes to encourage participants to work through the Course and apply the skills.
  Arms: Internet-based CBT intervention

SUMMARY:
Pain is the cardinal symptom of acute recurrent and chronic pancreatitis, and available medical treatments have limited efficacy. Pain self-management programs equip patients to minimize the impact of chronic painful conditions on activity, health, and psychosocial functioning. The purpose of the current study is to pilot the use of Internet-delivered pain self-management course in adults with chronic and acute recurrent pancreatitis to generate preliminary feasibility and acceptability data to inform design of a subsequent large randomized controlled trial.

DETAILED DESCRIPTION:
Acute recurrent pancreatitis (ARP) and chronic pancreatitis (CP) are associated with high disease burden across the lifespan. Recurring abdominal pain is the most prevalent and distressing symptom. Pain severity reduces health-related quality of life for individuals with CP and is associated with increased fatigue, anxiety and depressive symptoms, lower general health status, and reduced physical and role functioning. Medical therapies for CP pain have limited efficacy. Cognitive-behavioral interventions (CBT) offer safe and effective alternatives to pharmacological treatments for pain management. In other chronic painful conditions including gastrointestinal disorders, CBT interventions have been effective for reducing pain and pain impact including disability and depressive symptoms. CBT is traditionally provided by trained psychologists working with individual patients one-on-one or in small groups. Access to CBT is limited by availability of providers, with long waiting lists at centers offering CBT. The Internet is an ideal medium to provide pain self-management interventions that are low-cost and sustainable, and internet-based CBT has shown efficacy in children and adults with chronic pain, allowing clinics to greatly extend their reach to patients. The purpose of this study is to test the acceptability, feasibility, and preliminary efficacy of an Internet-delivered CBT pain self-management course for adults with acute recurrent and chronic pancreatitis pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Able and willing to provide informed consent for participation in this study
3. Meet CPDPC criteria for diagnosis of either suspected CP (CPDPC "yellow zone") or definite CP (CPDPC "red zone")
4. Have personal internet access on any device (e.g., phone, tablet, computer)
5. Has experienced pain intensity rated as 4 or higher on a 0-10 scale in the last month

Exclusion Criteria:

1. Currently undergoing treatment for cancer
2. Inability to understand English well enough to complete questionnaires or to participate in treatment
3. Severe depression (i.e., indicated by a score > 22 on the Patient Health Questionnaire (PHQ-9)
4. Significant suicidal ideation (i.e., indicated by a score > 2 to Question 9 of the PHQ-9)
5. Acutely suicidal or recent history of attempted suicide or self-harm (i.e., last 12 months)
6. Currently receiving treatment with a psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability | Immediately post-treatment
  Participants will complete a 12-item Treatment Evaluation Inventory questionnaire that assesses satisfaction and acceptability of the course of treatment and satisfaction with the outcome of the intervention. Items are rated on a 5-point Likert scale ranging from 1 = Strongly disagree, to 5 = Strongly agree.

SECONDARY OUTCOMES:
Treatment feasibility | Immediately post-treatment
  Feasibility will be determined by calculating rates of accrual, drop out, compliance, and missing data. Criteria for feasibility success will be based on: accrual rates >70%, attrition rates <15%, minimal technical difficulties (i.e., reported by <10%), adherence rates >80%, and minimal missing data.
Change in pain intensity | Baseline, 3-month follow-up
  Participants will report on presence and intensity of pain daily for 7 days at each assessment period. Pain intensity will be assessed using an 11-point numerical rating scale (NRS), where 0= no pain, and 10 = worst pain. Mean average intensity of the pain reported will serve as the pain measure.
Change in pain-related disability | Baseline, 3-month follow-up
  Participants will report their level of pain-related disability daily for 7 days at each assessment period. Questions of pain-related disability are taken from the Brief Pain Inventory and the Pain Disability Index. These measures assess the extent to which chronic pain disrupts aspects of daily life including social relations, work, mood, sleep, eating, and physical activity. All items are scored on a 0-10 NRS, with higher scores indicating greater disability.
Change in Disease specific and generic health related quality of life (HRQOL) | Baseline, 3-month follow-up
  Participants will complete the 18-item Pancreatitis Quality of Life Instrument to assess for disease-specific HRQOL difficulties. Items are scored on a 0-5 scale where 0 = Not applicable, 1 = Much less, and 5 = Much more. Participants will also complete the 12-item Short-Form Health Survey to assess for general HRQOL.
Change in Medication use | Baseline, 3-month follow-up
  Participants will record their medication use daily for 7 days at each assessment period
Change in Pain self-efficacy | Baseline, 3-month follow-up
  Participants will complete the 4-item Chronic Pain Self-Efficacy Scale. This scale assesses perceived self-efficacy over three factors: pain management, coping with symptoms, and physical function. All items are scored on a 7-point Likert scale where 0 = Not at all confident, and 6 = Completely confident
Change in Psychological distress | Baseline, 3-month follow-up
  Participants will complete the 4-item Anxiety and 4-item Depression subscales of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile to assess for levels of psychological distress over the past week. Items are scored on a 5-point Likert scale ranging from 1 = Never, to 5 = Always.
Change in Sleep and Fatigue | Baseline, 3-month follow-up
  Participants will complete the 4-item Sleep Disturbance and 4-item Fatigue subscales of the PROMIS-29 Profile to assess for problems with fatigue and sleep over the previous week. All items are scored on a 5-point Likert scale ranging 1 = Not at all, to 5 = Very much, except for one sleep item which is scored 1 = very poor, to 5 = Very good.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M Palermo, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palermo TM, Law EF, Topazian MD, Slack K, Dear BF, Ko YJ, Vege SS, Fogel E, Trikudanathan G, Andersen DK, Conwell DL, Yadav D; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). Internet Cognitive-Behavioral Therapy for Painful Chronic Pancreatitis: A Pilot Feasibility Randomized Controlled Trial. Clin Transl Gastroenterol. 2021 Jun 18;12(6):e00373. doi: 10.14309/ctg.0000000000000373. PMID 34140460
- [Derived] Yadav D, Palermo TM, Phillips AE, Bellin MD, Conwell DL. Painful chronic pancreatitis - new approaches for evaluation and management. Curr Opin Gastroenterol. 2021 Sep 1;37(5):504-511. doi: 10.1097/MOG.0000000000000769. PMID 34172622